CLINICAL TRIAL: NCT01076400
Title: A Two Part, Phase I-IIa Study Evaluating MK1775 in Combination With Topotecan/Cisplatin in Adult Patients With Cervical Cancer
Brief Title: A Study of Adavosertib (MK-1775) in Combination With Topotecan/Cisplatin in Participants With Cervical Cancer (MK-1775-008)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor permanently suspended new enrollment into the trial and discontinued the study; which was not related to any concerns over product safety.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1775-008; MK-1775-008 (Other: Merck Protocol Number); 2009-017054-12 (EudraCT Number)
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Results first posted 2017-12-14 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — adavosertib; Topotecan; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: adavosertib + topotecan/cisplatin (Experimental): Part 1: Dose escalation study. adavosertib capsules will be administered in sequentially rising dose levels twice daily for a total of nine doses on Days 1-5 of a 21-day cycle. Topotecan will be administered at a dosage of 0.75 mg/m^2 by intravenous (IV) infusion over 30 minutes on Days 1-3 . Cisplatin will be administered at a dosage of 50 mg/m^2 by IV infusion over 30 minutes on Day 1.
  Interventions: Drug: adavosertib; Drug: Topotecan; Drug: Cisplatin
- Part 2: adavosertib + topotecan/cisplatin (Experimental): Part 2: adavosertib capsules will be administered at the dose determined in Part 1 twice daily for a total of nine doses on Days 1-5 of a 21-day cycle. Topotecan will be administered at a dosage of 0.75 mg/m^2 by intravenous (IV) infusion over 30 minutes on Days 1-3. Cisplatin will be administered at a dosage of 50 mg/m^2 by IV infusion over 30 minutes on Day 1.
  Interventions: Drug: adavosertib; Drug: Topotecan; Drug: Cisplatin
- Part 2: Placebo to adavosertib + topotecan/cisplatin (Placebo Comparator): Part 2: Placebo to adavosertib capsules will be administered twice daily for a total of nine doses on Days 1-5 of a 21-day cycle. Topotecan will be administered at a dosage of 0.75 mg/m^2 by intravenous (IV) infusion over 30 minutes on Days 1-3. Cisplatin will be administered at a dosage of 50 mg/m^2 by IV infusion over 30 minutes on Day 1.
  Interventions: Drug: Topotecan; Drug: Cisplatin; Drug: Placebo to adavosertib

INTERVENTIONS:
Drug: adavosertib — Adavosertib capsules are administered in sequentially rising dose levels twice daily for a total of nine doses on Days 1-5 of a 21-day cycle.
  Other Names: MK-1775
  Arms: Part 1: adavosertib + topotecan/cisplatin; Part 2: adavosertib + topotecan/cisplatin
Drug: Topotecan — Topotecan is administered at a dosage of 0.75 mg/m^2 by intravenous (IV) infusion over 30 minutes on Days 1-3.
Drug: Cisplatin — Cisplatin is administered at a dosage of 50 mg/m^2 by IV infusion over 30 minutes on Day 1.
Drug: Placebo to adavosertib — Placebo to adavosertib capsules are administered in sequentially rising dose levels twice daily for a total of nine doses on Days 1-5 of a 21-day cycle.
  Arms: Part 2: Placebo to adavosertib + topotecan/cisplatin

SUMMARY:
This study will be conducted in two parts. Part 1 will determine whether administration of adavosertib in combination with topotecan and cisplatin is generally well-tolerated and causes clinical objective responses in patients with cervical cancer. Part 1 will also define the recommended Phase 2 dose and maximum tolerated dose (MTD) of the combination of adavosertib with topotecan and cisplatin. Part 2 of the study will evaluate whether treatment with adavosertib in combination with topotecan and cisplatin causes an improvement in progression-free survival (PFS) compared to treatment with topotecan and cisplatin alone and will further evaluate the tolerability of the combination treatment. The primary hypothesis is the combination of adavosertib, topotecan and cisplatin causes objective radiological responses (assessed per Response Evaluation Criteria in Solid Tumors [RECIST] 1.1 criteria) in ≥30% of participants. Due to the early termination of the study by the sponsor, no participants were enrolled in Part 2 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Has advanced, metastatic, and recurrent squamous cell, adenosquamous, or adeno-carcinoma of the uterine cervix (Stage II - IVb)
* Has received cisplatin in combination with radiation as initial or adjuvant treatment for their cervical cancer
* Has not received any other treatment for their cancer following the cisplatin-based chemo-radiation or targeted therapy except non-cytotoxic targeted therapy
* Recurrence must be at least 6 months post cisplatin-based chemotherapy
* Has measurable disease
* Performance status on the Eastern Cooperative Oncology Group (ECOG) Performance Scale is less than or equal to 1
* Has a negative pregnancy test within 72 hours of the first dose of study medication

Exclusion Criteria:

* Has had chemotherapy, radiotherapy, or biological therapy within 6 months of entering the study
* Has a history of vascular thrombotic events or vascular reconstruction
* Has active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has a primary CNS tumor
* Requires the use of medications or products that are metabolized by, or inhibit or induce CYP3A4 (Cytochrome P450 3A4)
* Is expecting to reproduce within the duration of the study or is pregnant or breastfeeding
* Is known to be Human Immunodeficiency Virus (HIV)-positive
* Has known active Hepatitis B or C
* Has a known history of interstitial lung disease or pulmonary fibrosis
* Has symptomatic ascites or pleural effusion
* Has a clinical history suggestive of Li-Fraumeni Syndrome

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 7 (Actual)
Dates: Start 2010-05-31 (Actual); Primary Completion 2011-06-13 (Actual); Study Completion 2011-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trial Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Due to the early termination of the study by the sponsor, no participants were enrolled in Part 2 of the study.
Groups:
- Part 1: MK-1775 + Topotecan/Cisplatin: Part 1: MK-1775 capsules were administered at 50 mg twice daily on Days 1-4, and once on Day 5 for a total of nine doses per cycle. Each cycle was 21 days. Topotecan was administered at a dosage of 0.75 mg/m^2 by intravenous (IV) infusion over 30 minutes on Days 1-3 of each cycle. Cisplatin was administered at a dosage of 50 mg/m^2 by IV infusion over 30 minutes on Day 1 of each cycle. Only a single dose of MK-1775 was administered during Part 1.
- Part 2: MK-1775 + Topotecan/Cisplatin: Part 2: MK-1775 capsules will be administered at the dose determined in Part 1 twice daily for a total of nine doses on Days 1-5 of a 21-day cycle. Topotecan will be administered at a dosage of 0.75 mg/m^2 by intravenous (IV) infusion over 30 minutes on Days 1-3. Cisplatin will be administered at a dosage of 50 mg/m^2 by IV infusion over 30 minutes on Day 1.
- Part 2: Placebo to MK-1775 + Topotecan/Cisplatin: Part 2: Placebo to MK-1775 capsules will be administered twice daily for a total of nine doses on Days 1-5 of a 21-day cycle. Topotecan will be administered at a dosage of 0.75 mg/m^2 by intravenous (IV) infusion over 30 minutes on Days 1-3. Cisplatin will be administered at a dosage of 50 mg/m^2 by IV infusion over 30 minutes on Day 1.
Period: Overall Study
Arm/Group | Part 1: MK-1775 + Topotecan/Cisplatin | Part 2: MK-1775 + Topotecan/Cisplatin | Part 2: Placebo to MK-1775 + Topotecan/Cisplatin
Started | 7 | 0 (No participants were enrolled in Part 2 of the study.) | 0 (No participants were enrolled in Part 2 of the study.)
Completed | 0 | 0 | 0
Not Completed | 7 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Progressive Disease | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Part 1: MK-1775 + Topotecan/Cisplatin
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.3 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Percentage of Participants Whose Best Confirmed Response is Partial Response (PR) or Complete Response (CR)
Description: On the basis of Response Evaluation Criteria In Solid Tumors (RECIST) 1.1, PR is at least a 30% decrease in the sum of the longest diameters (SLD) of target lesions, taking as reference the baseline sum diameters. CR is the disappearance of all extranodal target lesions, where all pathological lymph nodes must have decreased to <10 mm in the short axis.
Time Frame: Up to approximately 1 year
Population: The study was prematurely terminated, and data were not collected, so no analyses were performed.
Arm/Group | Part 1: MK-1775 + Topotecan/Cisplatin
Number analyzed (Participants) | 0

2. Primary Outcome: Part 1: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: A DLT is a protocol-defined, (hematologic and non-hematologic), AE that must be definitely, probably, or possibly related to the study therapy. A DLT is any of the following: Grade 4-5 hematological toxicity; Grade 3 or Grade 4 neutropenia with fever >38.°C and/or infection requiring antibiotic or anti-fungal treatment. Non-hematologic dose-limiting toxicities are any Grade 3, 4, or 5 non-hematologic toxicity, with specific exceptions. If occurring within the first cycle of combination therapy: unresolved drug-related toxicity, preventing (re) treatment for 3 weeks or more from the date of the next scheduled treatment or any drug-related toxicity preventing the participant from taking at least 75% of the doses of MK-1775 with each administration of chemotherapy.
Time Frame: Up to approximately 1 year
Population: Participants who completed the first cycle of combination therapy or discontinued from the study due to a DLT attributable to study therapy. One participant who violated the protocol was not assessed for DLTs.
Measure: Number; unit: Number of participants
Arm/Group | Part 1: MK-1775 + Topotecan/Cisplatin
Number analyzed (Participants) | 6
Number of participants | 2

3. Primary Outcome: Part 2: Length of Time for Progression-free Survival (PFS)
Description: PFS is the length of time during and after treatment that a participant lives, but whose tumor progression does not worsen. PFS is defined as the time from randomization to progressive disease or death, whichever occurs earlier. Tumor volume changes of +20% for progressive disease was used to be consistent with RECIST 1.1.
Time Frame: Up to approximately 1 year
Population: Due to the early termination of the study Part 2 was not performed.
Arm/Group | Part 1: MK-1775 + Topotecan/Cisplatin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: At least 30 days following last dose of study therapy or until death (up to approximately 1 year).
Description: All randomized participants who received at least one dose of study treatment.
Arm/Group | Part 1: MK-1775 + Topotecan/Cisplatin
Serious Adverse Events (participants affected / at risk) | 5/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: MK-1775 + Topotecan/Cisplatin (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: MK-1775 + Topotecan/Cisplatin (N=7)
Anaemia (Blood and lymphatic system disorders) | 6 (17)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 6 (18)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (19)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Constipation (Gastrointestinal disorders) | 4 (7)
Diarrhoea (Gastrointestinal disorders) | 4 (5)
Dyspepsia (Gastrointestinal disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (9)
Vomiting (Gastrointestinal disorders) | 3 (10)
Asthenia (General disorders) | 4 (7)
Chest pain (General disorders) | 1 (1)
Discomfort (General disorders) | 1 (3)
Fatigue (General disorders) | 2 (5)
Influenza like illness (General disorders) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (2)
Rhinitis (Infections and infestations) | 1 (2)
Skin infection (Infections and infestations) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 1 (5)
Blood magnesium decreased (Investigations) | 1 (1)
Blood sodium decreased (Investigations) | 1 (4)
Haemoglobin decreased (Investigations) | 1 (4)
Neutrophil count decreased (Investigations) | 2 (3)
Platelet count decreased (Investigations) | 1 (3)
Weight decreased (Investigations) | 1 (1)
White blood cell count decreased (Investigations) | 2 (5)
Decreased appetite (Metabolism and nutrition disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (6)
Lethargy (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (2)
Pelvic venous thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission.